CLINICAL TRIAL: NCT07040059
Title: A Phase 1b/2, Open-label, Randomized, Multicenter Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of AUR103 Calcium in Patients With HER2-positive Advanced Gastric/Gastroesophageal Junction Adenocarcinoma (BHARAT-2)
Brief Title: A Phase 1b/2 Clinical Trial Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of AUR103 Calcium in Patients With HER2-positive Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUR103-201
Record Dates: First submitted 2025-06-04; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HER 2 Positive Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: BHARAT 2
MeSH Terms: interventions — Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: The Phase 1 of the study is a single-arm study, which will be conducted in a dose-escalation manner by following 3 + 3 traditional design. The Phase 2 of the study is a randomized study with either two or three groups with parallel study design. The number of groups in the Phase 2 part of the study will be decided based on the safety, PK and/or PD data from Phase 1.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b (Cohort 1: AUR103 Calcium 200 mg BID with standard dose of Trastuzumab and CAPOX. (Experimental): Phase 1b: Cohort 2 (AUR103 Calcium 300 mg BID with standard dose of Trastuzumab and CAPOX). Cohort 2 of Phase 1b will start after completion of dose-limiting toxicity (DLT) period of Cohort 1.
  Interventions: Drug: AUR103 Calcium
- Phase 2 Treatment Arm (Experimental): Phase 2 (Experimental Arm) - Either one or two treatment arm(s) selected from the Phase 1b part.
  Interventions: Drug: AUR103 Calcium
- Phase 2 Control Arm (Active Comparator): Phase 2 will have control arm (with standard dose of Trastuzumab and CAPOX).
  Interventions: Drug: Trastuzumab + CAPOX (Capecitabine + Oxaliplatin)
- Phase 1b (Cohort 2: AUR103 Calcium 300 mg BID with standard dose of Trastuzumab and CAPOX. (Experimental)
  Interventions: Drug: AUR103 Calcium
- Phase 1b: Cohort 3 (AUR103 Calcium 400 mg BID with standard dose of Trastuzumab and CAPOX). (Experimental): Phase 1b: Cohort 3 (AUR103 Calcium 400 mg BID with standard dose of Trastuzumab and CAPOX). Cohort 3 of Phase 1b will start after completion of dose-limiting toxicity (DLT) period of Cohort 2.
  Interventions: Drug: AUR103 Calcium

INTERVENTIONS:
Drug: AUR103 Calcium — AUR103 Calcium will be administered with standard dose of Trastuzumab and CAPOX (Capecitabine and oxaliplatin).
  Other Names: Trastuzumab; Capecitabine
  Arms: Phase 1b (Cohort 1: AUR103 Calcium 200 mg BID with standard dose of Trastuzumab and CAPOX.; Phase 1b (Cohort 2: AUR103 Calcium 300 mg BID with standard dose of Trastuzumab and CAPOX.; Phase 1b: Cohort 3 (AUR103 Calcium 400 mg BID with standard dose of Trastuzumab and CAPOX).; Phase 2 Treatment Arm
Drug: Trastuzumab + CAPOX (Capecitabine + Oxaliplatin) — Standard dose of Trastuzumab and CAPOX (Capecitabine + Oxaliplatin) will be administered in the Control Arm of Phase 2.
  Other Names: Trastuzumab; Capecitabine
  Arms: Phase 2 Control Arm

SUMMARY:
The study will have a dose escalation part (Phase 1b) and a randomized part (Phase 2). In Phase 1b, patients diagnosed with advanced HER2 positive gastric/gastroesophageal adenocarcinoma will be enrolled in a 3 + 3 design dose escalation manner to evaluate the safety, efficacy, PK/PD of AUR103 Calcium when administered in combination with Trastuzumab and CAPOX (capecitabine and oxaliplatin). Phase 2 is a randomization study. The primary objective of the phase 2 study is to assess the efficacy of AUR103 Calcium when administered in combination with Trastuzumab and CAPOX (capecitabine and oxaliplatin). The phase 2 of the study will be conducted after Phase 1b.

DETAILED DESCRIPTION:
This study (AUR103-201; BHARAT-2) will be conducted in patients with HER2-positive gastric or gastroesophageal (GE) junction adenocarcinoma, in the first-line setting. In the study Part 1 (Phase 1b), the safety and tolerability of AUR103 calcium will be evaluated in combination with Trastuzumab and CAPOX. In the study part 1 (Phase 1b), there will 3 cohorts; Cohort 1 patients will receive the study drug (AUR103 Calcium) at 200 mg BID dose along with standard doses of trastuzumab, and CAPOX (capecitabie and oxaliplatin), Cohort 2 patients will receive the study drug (AUR103 Calcium) at 300 mg BID dose along with standard doses of trastuzumab, and CAPOX, and Cohort 3 patients will receive the study drug (AUR103 Calcium) at 400 mg BID dose along with standard doses of trastuzumab, and CAPOX.

In the study Part 2 (Phase 2), the efficacy of AUR103 calcium in combination with Trastuzumab and CAPOX will be evaluated in HER2-positive gastric or gastroesophageal junction adenocarcinoma patients. The part 2 (Phase 2) of the study will be a randomized study which will start after part 1 (Phase 1b). In the study part 2 (Phase 2), there will either 1 or 2 treatment arm(s) and one control arm (Trastuzumab + CAPOX). The number treatment arms will be based on the phase 1b data. However, the treatment patients in the Phase 2 will receive the study drug along with Trastuzumab and CAPOX.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent and agree to comply with all study related activities.
2. Male or female patients aged greater than or equal to 18 years.
3. Patients must meet the following criteria for each of the respective parts of the study:

   a) Pathological diagnosis of a HER2-positive, unresectable locally advanced or metastatic, gastric / gastroesophageal (GE) junction adenocarcinoma.

   [Note: For patients who have already undergone HER2 testing, it does not need to be repeated. For patients who have not undergone HER2 testing, the same can be done as part of pre-screening, after taking informed consent].

   B) Patients must NOT have received any systemic anti-cancer therapy for the treatment of gastric or gastroesophageal (GE) junction adenocarcinoma.

   [Note: The partial resection of tumor or debulking surgery is allowed but any therapeutic chemotherapy or systemic anti-cancer therapy is not allowed].
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
5. Acceptable bone marrow as described below:

   1. ANC greater than or equal to 1500/μL (without WBC growth factor support).
   2. Platelet count greater than or equal to 100,000/μL (without transfusion support).
   3. Hemoglobin greater than or equal to 9 g/dL (Transfusion is allowed to achieve this Hb).
6. Acceptable organ function as described below:

   1. Total Bilirubin less than or equal to 1.5 x ULN (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin less than or equal to 2.5 x ULN).
   2. AST (SGOT) less than or equal to 3 x ULN (less than or equal to 5 × ULN if known liver metastases).
   3. ALT (SGPT) less than or equal to 3 x ULN (less than or equal to 5 × ULN if known liver metastases).
   4. Creatinine clearance (CrCl) greater than or equal to 60 mL/min (either measured or estimated by the Cockcroft-Gault formula). (Cockcroft-Gault formula for estimated creatinine clearance [eCrCl]: eCrCl = [140 - Age] × Weight [kg] × [0.85 if Female] / [72 × serum creatinine (mg/dL)]).
   5. Albumin greater than or equal to 3.0 g/dL.
7. Evidence of measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 [Note: Measurable disease for solid tumors is defined as at least one lesion that can be accurately measured in at least 1 dimension with a minimum size of 10 mm for non-nodal lesions or 15 mm in short axis for nodal lesions].
8. Patients who have not undergone HER2 testing must be willing and able to provide an adequate archived tumor tissue sample or a fresh tumor tissue sample to confirm HER2 status.

   [Note: If archived sample is not available, and HER2 testing has not been done, then patient must agree to submit fresh tumor sample for an assessment of HER2 status].
9. Left ventricular ejection fraction (LVEF) greater than or equal to 50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan at Screening.
10. Ability to swallow and retain oral medications.
11. Negative serum pregnancy test in women of childbearing potential (WOCBP).
12. Women of childbearing potential and men who partner with such a woman of childbearing potential must agree to use one or more of highly effective method(s) for contraception for the duration of the study, i.e., through 28-day follow up visit, after discontinuation of study drug(s).

Exclusion Criteria:

1. Patients with resectable gastric / gastroesophageal (GE) junction adenocarcinoma.
2. Exposed to definitive radiotherapy [Note: Palliative radiotherapy is allowed].
3. Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
4. Known central nervous system (CNS) metastases.
5. Major surgery less than or equal to 28 days from Cycle 1 Day 1 (Major surgery is defined as a procedure requiring general anaesthesia).
6. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness.
7. Known active or chronic hepatitis B or hepatitis C infection.
8. Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1.
9. Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in past 3 months, before Cycle 1 Day 1.
10. The QTcF (corrected QT interval Fridericia method) value in the screening ECG more than 460 ms in males and females.
11. Currently taking warfarin or other oral coumarin-derivative anticoagulant therapy.
12. Patients with peripheral neuropathy of Grade greater than or equal to 2.
13. Patients with severe obstructive pulmonary disease, pulmonary fibrosis, or interstitial lung disease.
14. Patients with poorly controlled hypertension, defined as systolic blood pressure more than or equal to 160 mmHg or diastolic blood pressure more than 100 mmHg.
15. Previous or concomitant additional malignancy, except for basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix; patients with other malignancies are eligible if they have remained disease free for at least 2 years prior to trial entry and in the opinion of the investigator deemed to have a low likelihood of recurrence.
16. Any clinically significant medical, psychiatric, or social condition; or laboratory abnormality that may increase the risk of trial participation or may interfere with the informed consent process and/or with compliance with the requirements of the trial or may interfere with the interpretation of the trial results and, in the Investigator's opinion, would make the patient inappropriate for entry into this trial.
17. Pregnant or lactating women.
18. Current swab-positive or suspected (under investigation) COVID19 infection or fever and other signs or symptoms suggestive of COVID-19 infection with recent contact of person(s) with confirmed COVID-19 infection, at screening or Cycle 1 Day 1.
19. Patients with any known contraindication to receive trastuzumab, or capecitabine, or oxaliplatin.
20. Known hypersensitivity to trastuzumab, capecitabine, oxaliplatin, or to any of its components.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Safety): Treatment Emergent Adverse Events (TEAEs) | Through the study completion, an average of 1 year
  TEAEs will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0)
Part 1 (Pharmacokinetics): Area under the curve (AUC) | On Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Area under the curve of AUR103 Calcium
Part 1 (Pharmacokinetics): Maximum concentration | On Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Maximum concentration of AUR103 Calcium
Part 1 (Pharmacokinetics): Time to Maximum concentration | On Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Time to Maximum concentration of AUR103 Calcium
Part 1 (Pharmacokinetics): Terminal elimination half life | On Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Terminal elimination half-life of AUR103 Calcium
Part 2 (Efficacy): Best Objective Tumor Response Rate (ORR) | Every 3 cycle, through study completion, for an average duration of one year.
  Best Objective Tumor Response Rate (ORR) will be assessed during the study

SECONDARY OUTCOMES:
Part 1 (Efficacy): Best Objective Tumor Response Rate (ORR) | Every 3 cycle, through study completion, for an average duration of one year.
  ORR will be assessed during the study during the study
Part 1 (Efficacy): Duration of response (DoR) | Every 3 cycle, through study completion, for an average duration of one year.
  Duration of response (DoR) will be assessed during the study
Part 1 (Efficacy): Time to Objective Tumor Response | Every 3 cycle, through study completion, for an average duration of one year.
  Time to Objective Tumor Response will be assessed during the study
Part 1 (Efficacy): Duration of Clinical Benefit Rate (CBR) | Every 3 cycle, through study completion, for an average duration of one year.
  Duration of Clinical Benefit Rate (CBR) will be assessed during the study
Part 1 (Efficacy): Clinical Benefit Rate (CBR) | Every 3 cycle, through study completion, for an average duration of one year.
  Clinical Benefit Rate (CBR) will be assessed during the study
Part 1 (Efficacy): Progression Free Survival (PFS) | Every 3 cycle, through study completion, for an average duration of one year.
  Progression Free Survival (PFS) will be assessed during the study
Part 1 (Efficacy): Time to progression | Every 3 cycle, through study completion, for an average duration of one year.
  Time to progression will be assessed during the study
Part 1 (Efficacy): Overall survival (OS) | Through study completion, an average of 1 year
  Overall survival will be assessed during the study
Part 2 (Efficacy): Duration of response | Every 3 cycle, through study completion, for an average duration of one year.
  Duration of response will be assessed during the study
Part 2 (Efficacy): Time to Objective Tumor Response | Every 3 cycle, through study completion, for an average duration of one year.
  Time to Objective Tumor Response will be assessed during the study
Part 2 (Efficacy): Clinical Benefit Rate (CBR) | Every 3 cycle, through study completion, for an average duration of one year.
  Clinical Benefit Rate (CBR) will be assessed during the study
Part 2 (Efficacy): Duration of Clinical Benefit Rate (CBR) | Every 3 cycle, through study completion, for an average duration of one year.
  Duration of Clinical Benefit Rate (CBR) will be assessed during the study
Part 2 (Efficacy): Progression Free Survival (PFS) | Every 3 cycle, through study completion, for an average duration of one year.
  Progression Free Survival (PFS) will be assessed during the study
Part 2 (Efficacy): Time to progression | Every 3 cycle, through study completion, for an average duration of one year.
  Time to progression will be assessed during the study
Part 2 (Efficacy): Overall survival (OS) | Through study completion, an average of 1 year
  Overall survival will be assessed during the study
Part 2 (Safety): Treatment Emergent Adverse Events (TEAEs) | Through study completion, an average of 1 year
  Treatment Emergent Adverse Events (TEAEs) will be assessed throughout the study duration
Part 2 (Health Related Quality of Life): EORTC QLQ-C30 | Cycle 1 Day 1 and Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Health Related Quality of Life will be assessed by EORTC QLQ-C30 questionaire
Part 2 (Health Related Quality of Life): EORTC-QLQ-STO22 score | Cycle 1 Day 1 and Day 1 of each subsequent cycle through study completion, for an average duration of one year.
  Health Related Quality of Life will be assessed by EORTC-QLQ-STO22 score

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Kumar, Principal Investigator — Aurigene Oncology Limited
Locations (8):
- India (8):
  - HCG Cancer Center, Vizag, Andhra Pradesh
  - Shalby Hospital, Ahmedabad, Gujarat
  - The Gujarat Cancer & Research Insititute, Ahmedabad, Gujarat
  - Kiran Hospital Multi Super Speciality Hospital & Reseach Center, Surat, Gujarat
  - Asha Hospital and Research Centre, Bangalore, Karnataka
  - Karnataka Cancer Hospital and Radiation Theraphy Center, Bangalore, Karnataka
  - Netaji Subhas Chandra Bose Cancer Hospital, Kolkata, West Bengal
  - Hope & Heal Cancer Hospital and Research Center, Siliguri, West Bengal

IPD SHARING:
Plan to Share IPD: No
Due to ethical concerns.